CLINICAL TRIAL: NCT06423729
Title: Clinical Study Evaluating the Effect of Nicorandil in Type 2 Diabetic Obese Patients Treated With Sulfonylurea
Brief Title: Effect of Nicorandil in Type 2 Diabetic Obese Patients
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Merna Mohamed Seddik Ali, Merna Mohamed Seddik Ali , Master degree in Clinical Pharmacy, Tanta University, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nicorandil in DM
Record Dates: First submitted 2024-05-16; First posted 2024-05-21 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 DM, Nicorandil, Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Nicorandil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): 23 patients who will receive 2nd generation sulfonylureas only, for three months.
- Nicorandil Arm (Experimental): 23 patients who will receive a combination of 2nd generation sulfonylureas and nicorandil 10 mg twice daily,for three months.
  Interventions: Drug: Nicorandil 10 MG

INTERVENTIONS:
Drug: Nicorandil 10 MG — Patients will receive oral Nicorandil 10 MG twice daily in addition to 2nd generation sulfonylureas , for 3 months.
  Arms: Nicorandil Arm

SUMMARY:
1. Evaluating the effect of nicorandil on glycemic control of diabetic obese patients treated with sulfonylureas.
2. Investigating the effect of nicorandil on body weight of diabetic obese patients treated with sulfonylureas.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes duration ranged from 1 to 10 years.
* Body mass index (BMI) >30 Kg/m2.
* The selected patients are treated with sulfonylureas alone.
* The age of selected patient ranged from 18 and 60 years.

Exclusion Criteria:

* Pregnant and lactating females.
* Patients with hypersensitivity to nicorandil.
* Uncontrolled hypertension and its antihypertensive medications
* Severe renal or hepatic disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c level | The participants will be assessed before initiation of the study (baseline), and at the end of the study after 3 months.
  Change in HbA1c (From baseline to 12 weeks)
Change in body weight. | The participants will be assessed before initiation of the study (baseline), and at the end of the study after 3 months.
  Change in body weight (From baseline to 12 weeks).
Change in Body mass index (BMI) | The participants will be assessed before initiation of the study (baseline), and at the end of the study after 3 months.
  Change in Body mass index (BMI) (From baseline to 12 weeks).
Change in Visceral adiposity index (VAI). | The participants will be assessed before initiation of the study (baseline), and at the end of the study after 3 months.
  Change in Visceral adiposity index (VAI) (From baseline to 12 weeks).

SECONDARY OUTCOMES:
Change in Adiponenctin, Interleukin-6 (IL-6) and Nitric oxide (NO) serum levels. | The participants will be assessed before initiation of the study (baseline), and at the end of the study after 3 months.
  Assessment of Adiponenctin, Interleukin-6 (IL-6) and Nitric oxide levels by ELISA Kits according to manufacturer's instructions.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pharmacy, Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No